CLINICAL TRIAL: NCT05714280
Title: Developing a Tailored, Theoretically-Driven Smartphone Physical Activity Intervention for African American Women
Brief Title: PA4Health Physical Activity App Open Pilot Study for African American Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CityUNYSPH; K23MD014164 (NIH)
Record Dates: First submitted 2022-06-28; First posted 2023-02-06 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Test Acceptability/Usability of a Physical Activity App Developed for African American Women
Keywords: PA4Health Open Pilot; Physical Activity App; African American Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: PA4Health Open Pilot — The goal of this aim is to collect data that guide the refinement of intervention components and structure to increase appeal to AA women. Fifteen physically inactive AA women will participate in a 12-week study examining the feasibility, acceptability, and usage of the PA4Health app.
  They will receive a Fitbit tracker to be worn during the trial. Following the trial, participants will complete self-report measures as well as a semi-structured interview to learn about their experience in using the app, any experienced difficulties, and recommendations for improving the acceptance and usage of the app.

SUMMARY:
Test the acceptability of a smartphone physical activity app for African American women

DETAILED DESCRIPTION:
The goal of this aim is to collect data that guide the refinement of intervention components and structure to increase appeal to AA women. Fifteen physically inactive AA women will participate in a 12-week study examining the feasibility, acceptability, and usage of the PA4Health app. They will receive a Fitbit tracker to be worn during the trial. Following the trial, participants will complete self-report measures as well as a semi-structured interview to learn about their experience in using the app, any experienced difficulties, and recommendations for improving the acceptance and usage of the app.

Intervention components: The intervention components include: tailored daily text intervention text message, educational feature, goal setting and monitoring, and an activity locator that allow participants to enter their zip code and view available resources for physical activity.

ELIGIBILITY:
Inclusion: Eligible participants must:

1. be ages 18-64
2. identify as AA and female
3. own a smartphone
4. be able to provide consent
5. not regularly physically active (i.e. less than 90 mins. of MVPA per week), 6) medically cleared for PA,

7) have a valid email address, and 9) no previous engagement in the study.

Exclusion: Individuals will be excluded if they report:

1. physical limitations to PA engagement
2. significant medical conditions (e.g., heart failure)
3. planned surgery in the next 6 months,
4. pregnant or plan to become pregnant in the next 6 months.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
System usability scale (SUS)-- app satisfaction | 8 weeks study
  The SUS measures ability of technology software. High levels of usability and acceptability of the app will be determined by a score greater than 70 on the SUS. Information will be used for improvement of the software.
Metada; collected through app system | 8weeks
  This information will inform usage of patterns of participants, including how frequently the logged into the app system and the component of the app the more frequently or less frequently

SECONDARY OUTCOMES:
Accelerometer | Participants will wear this device for 7 consecutive days at baseline and at 8 weeks(end of the intervention)
  actigraph data will be analyzed to explore potential changes over time objectively collected min/week of MVPA
Fitbit data | Participants will wear this device daily during the 8-week intervention
  Fitbit data will be explored to estimate the effect of the intervention on mean steps/week over time

CONTACTS AND LOCATIONS:
Locations (1):
- City University of New York School of Public Health & Health Policy, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No